CLINICAL TRIAL: NCT06629376
Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Pharmacological Studies of SSS11 in Patients With Gout and Hyperuricemia After Multiple Administrations, Dose Escalation, Randomized Double-blind, Placebo-controlled Trials
Brief Title: Safety, Tolerability, and Pharmacokinetic Characteristics of SSS11 in Patients With Gout and Hyperuricemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSS-SSS11-UND-I-03
Record Dates: First submitted 2024-09-06; First posted 2024-10-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-10

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Experimental： group1 (Experimental): injection；strength；4mg
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection
- Experimental： group2 (Experimental): injection；strength；8mg
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection
- Experimental： group3 (Experimental): injection；strength；12mg
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection
- Experimental： group4 (Experimental): injection；strength；16mg
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection
- Experimental： group5 (Experimental): injection；strength；20mg
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection
- Placebo control group (Placebo Comparator): The same volume of placebo as SSS11
  Interventions: Drug: Pegylated Recombinant Candida Utilis Uricase for Injection

INTERVENTIONS:
Drug: Pegylated Recombinant Candida Utilis Uricase for Injection — According to the dosage requirements of each experimental group, intravenous infusion should be administered for at least 2 hours each time
  Other Names: SSS11

SUMMARY:
This is a safety, tolerability, pharmacokinetics, and preliminary pharmacological study of multiple administration, dose escalation, randomized double-blind, placebo-controlled.The main purpose of this experiment is to evaluate the safety and tolerability of multiple injections of PEGylated recombinant Candida urate oxidase (test drug code: SSS11) in patients with gout and hyperuricemia.The experimental period includes a screening period of 4 weeks, a treatment period of 4 or 8 weeks, and an observation period of 4 weeks。

ELIGIBILITY:
Inclusion Criteria:

* A patient with clinical diagnosis of gout (according to the 2015 ACR/EULAR gout classification criteria), non acute attack phase, and hyperuricemia {under normal purine diet, blood uric acid>420 µ mol/L (7 mg/dl) not tested twice on an empty stomach on the same day}。
* Screening period blood uric acid>420 µ mol/L (7mg/dl)。

Exclusion Criteria:

* Within 14 days prior to enrollment (or within 5 half lives of the drug, whichever is longer), medication that lowers uric acid levels or affects uric acid levels and related drugs (allopurinol, febuxostat, benzbromarone, probenecid, benzenesulfonazolone, Tongyifengning tablets, etc.) must be taken, or during the study period, other drugs that lower uric acid levels or affect uric acid levels and related drugs other than experimental drugs must not be discontinued。
* Patients with acute gout attacks within 14 days prior to enrollment。
* Previously received uric acid oxidase or treated with similar drugs such as pegolase or rabulidase。
* Individuals with a history of glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD enzyme activity levels below the lower limit of normal。
* Individuals with a history of catalase deficiency or evidence that meets the diagnostic criteria for catalase deficiency。
* Malignant tumor patients (whether treated or not)。

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was safety. | up to 12 weeks
  Assessment AEs by frequency and severity

SECONDARY OUTCOMES:
Difference between post administration blood uric acid and baseline | up to 12 weeks
Duration of blood uric acid<360 μ mol/L | up to 12 weeks
Proportion of subjects with blood uric acid levels below 360 μ mol/L at each sample collection time point | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- HuaShan Hospital Fudan University project, ShangHai, China, Shanghai, China